CLINICAL TRIAL: NCT05026294
Title: Effects of Plyometric Exercises Versus Flatfoot Corrective Exercises on Postural Control and Foot Posture in Obese Children With Flexible Flatfoot
Brief Title: Plyometric Exercise With Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hatem Allam, Assistant professor, Taif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAP-02-T-067- 452
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Flat Feet
MeSH Terms: conditions — Flatfoot | interventions — Plyometric Exercise; Exercise

STUDY DESIGN:
Intervention Model Description: A Pretest-posttest control group design was used. A sample of 47 male children participated in the current study. After gathering the baseline measurements, the participants were randomly assigned into three groups: experimental group I, (EGI) contained 16 participants, experimental group II (EGII) contained 16 participants, and control group, (CG) contained 15. The stratification was done using sealed envelopes. The children were not aware of their group.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group I (Experimental): The experimental group received plyometric training
  Interventions: Other: plyometric exercises
- Experimental group II (Experimental): The experimental group received flat feet rehabilitation training
  Interventions: Other: Exercises for flat feet rehabilitation
- Control group (No Intervention): The Control group didn't receive intervention

INTERVENTIONS:
Other: plyometric exercises — Exercises for strength and flexibility
  Arms: Experimental group I
Other: Exercises for flat feet rehabilitation — Exercises for intrinsic muscles strength
  Arms: Experimental group II

SUMMARY:
Obesity is one of the main factors that contribute to an acquired flat foot deformity which in turn impairs the balance strategies. The purpose of the current study was to compare the effect of plyometric exercises with flatfoot corrective exercise on balance, foot posture, and functional mobility in obese children with flexible flatfoot.

DETAILED DESCRIPTION:
A sample of 47 male children participated in the current study. The participants were selected from different elementary schools in Taif, Saudi Arabia. Their age ranged from 7 to 11 years. the sample was randomly divided into 3 groups: the experimental group I, (EGI), the experimental group II, (EGII), and the control group (CG). The EGI received a plyometric exercise program. The EGII received the corrective exercises 2 sessions per week for 10 weeks. The control group did not perform any planned physical activities during the intervention period but continued in their routine physical activities. The Prokin system was used to assess the static balance, timed up and go test was used to assess functional mobility, and Navicular drop test was used to assess the degree of flatfoot deformity, prior to and after the intervention for all groups.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index percentile equal to or greater than the 95th percentile
* All had no previous history of strength or balance training or involvement in competitive sports emphasizing muscular strength or balance.
* All participants had balance deficiency and mobile flat foot.

Exclusion Criteria:

* Previous injury to the lower limb required medical care.
* Confounding conditions, such as a deformity of or surgery in the lower limb.
* visual impairment, or neuromuscular disorders.
* engagement in obesity treatment programs, three months prior to the study.

Ages: 7 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — A sample of 47 male children participated in the current study without having female participants because of the cultural perspective.
Enrollment: 47 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Foot posture | 10 weeks
  condition of the medial longitudinal arch of the foot
Balance (measure 1) | 10 weeks
  Perimeter area (mm).
Balance (measure 2) | 10 weeks
  Ellipse area (mm2).
Balance (measure 3) | 10 weeks
  Standard backward-forward deviation.
Balance (measure 4) | 10 weeks
  Standard medial-lateral deviation.
Functional mobility | 10 weeks
  Timed up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Allam, A.professor, Principal Investigator — Taif University
Locations (1):
- College of Applied Medical Sciences, Ta'if, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No